CLINICAL TRIAL: NCT05511948
Title: A Randomized, Observer-Blinded, Vehicle-Controlled Study on the Safety and Efficacy of Twice Daily Application of Ruboxistaurin (DBI-102) Gel Vs.Vehicle Gel Vs. Hydroquinone Cream on Sun-Exposed and Sun-Protected Skin of Adults
Brief Title: Randomized and Open Label Study for Safety and Efficacy of DBI-102 vs. Vehicle vs. Hydroquinone on Skin Pigmentation and Lentigos
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DermBiont, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: CT-212
Record Dates: First submitted 2022-08-20; First posted 2022-08-23 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Hyperpigmentation
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Intervention Model Description: Randomized 3-arm tranche of main cohorts, to be followed by open-label Solar Lentigo sub-cohort
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The open label sub-cohort will not have masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DBI-102 (Experimental): Topical DBI-102 Gel, 0.8% twice daily for 12 weeks for the randomized cohort
  Interventions: Drug: DBI-102
- Vehicle gel (Placebo Comparator): Inactive comparator
  Interventions: Drug: Vehicle gel
- Hydroquinone cream (Active Comparator): 4% Hydroquinone cream, Acella (approved), twice daily for 12 weeks
  Interventions: Drug: Hydroquinone Cream

INTERVENTIONS:
Drug: DBI-102 — Topical application on dorsal hand and upper volar arm
  Arms: DBI-102
Drug: Vehicle gel — Inactive comparator
  Arms: Vehicle gel
Drug: Hydroquinone Cream — 4% Hydroquinone cream, Acella (approved), twice daily for 12 weeks
  Arms: Hydroquinone cream

SUMMARY:
This is a randomized, observer-blinded, vehicle-controlled multi-dose trial that examines the effect of twice daily application of 0.8% DBI-102 Gel, 4% Hydroquinone cream, and Vehicle Gel for 12 weeks in adults with Fitzpatrick Skin Types IV-V and a colorimeter L* measurement between 57.8 and 46.1.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female at least 18 years of age.
* Must be Fitzpatrick Skin Type IV-V and have an L* measurement between 57.8 and 46.1, using the Chromometer CM-700.
* Ability to understand, agree to, and sign the study informed consent form (ICF).
* Agree to discontinue all agents used to treat hyperpigmentation, aging or exfoliate the skin during the course of the study. Makeup and moisturizers are permitted.
* Agree not to change their sun exposure at work, home, or leisure.
* Technical ability and willingness to apply test articles.
* Willing to allow digital photos of treatment and comparison areas to be taken and stored.

Additional Inclusion Criterion for the solar lentigo Sub-Cohort:

* At least 4 solar lentigos at least 4 mm in diameter present on each dorsal hand.

Exclusion Criteria:

* Positive urine pregnancy test, pregnant, lactating, or female of childbearing potential who does not agree to use an active method of birth control for the duration of the study.
* Conditions at baseline that would interfere with evaluation of UV-tanned skin, especially other pigmentary disorders including, but not limited to, melasma or vitiligo affecting the treatment and comparison sites.
* Presence of known concomitant diseases associated with the development of hyperpigmentation (e.g., thyroid, liver, adrenal).
* Current tanning booth exposure or any kind of phototherapy within 3 months of Screening.
* Current or past use of monobenzyl ether or hydroquinone (Benoquin) to depigment the skin.
* Past or recent use of any skin bleaching treatment within 6 months of Screening.
* A chemical peel within 3 months of Screening.
* Laser or light-based treatment of the treatment areas within 3 months of Screening.
* Use of any photosensitizing medications within the past 6 months of Screening, including psoralens, sulfonamide drugs, tetracycline antibiotics, thiazide diuretics, phenothiazines, coal tar and derivatives, and tricyclic antidepressants.
* Any dermatological conditions that could interfere with clinical evaluations or any disease state or physical condition which might expose the subject to an unacceptable risk by study participation.
* Any underlying disease(s) or other dermatological conditions that require the use of exclusionary topical or systemic therapy (see Exclusion criteria 5 and 6).
* Unwilling to discontinue applying any prescription or over the counter (OTC) topical product creams and ointments, other than makeup and moisturizers, on treatment area(s) at Baseline through their last day of study.
* Treatment of any type of cancer within 6 months of Screening with the exception of superficial skin cancers such as basal cell or squamous cell carcinoma.
* Known allergy to any of the test article(s) or any components in the test article(s) or history of hypersensitivity or allergic reactions to any of the study preparations as described in the Investigator's Brochure.
* History of active atopic dermatitis, as diagnosed by a physician, requiring treatment within the past 2 years.
* Unable to meet the study attendance requirements.
* Any history of psychiatric disease or history of alcohol or drug abuse that would interfere with the ability to comply with the study protocol.
* Participation in any other trial of an investigational drug or device within 30 days prior to enrollment or participation in a research study concurrent with this study.

Additional Exclusion Criterion for the Sub-Cohort

* Any previous treatment for solar lentigos on the dorsal hands.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-03-07 (Actual)

PRIMARY OUTCOMES:
Decrease in pigmentation based on melanin index | 12 weeks after first dose
  Change in L* and ITA colorimetry measurements
Decrease in pigmentation based on digital imaging | 12 weeks after first dose
  Change as measured with Canfield RBX software analysis

SECONDARY OUTCOMES:
Percent Change in Investigator Dynamic Grading Assessment (IDGA) | At weeks 2,4,6,8,10, and 12
  Percent pigmentation differences between treated and contralateral Percent Change in Investigator Dynamic Grading Assessment (IDGA)
Proportion of subjects with Improved Investigator Dynamic Grading Scale (IDGA) | At weeks 2,4,6,8,10, and 12
  Proportion of subjects with less pigmentation at treated sites vs contralateral untreated sites

CONTACTS AND LOCATIONS:
Overall Officials: David Zepeda, MD, Principal Investigator — Zepeda Dermatologia
Locations (1):
- Zepeda Dermatologia, Santa Tecla, La Libertad Department, El Salvador

IPD SHARING:
Plan to Share IPD: No